CLINICAL TRIAL: NCT05599048
Title: A Phase I/II Study of Hyperpolarized 13C MRI as a Biomarker of Aggressiveness & Response to Therapy in Patients With Advanced Solid Tumors
Brief Title: Hyperpolarized 13C MRI as a Biomarker in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Robert Bok, MD, PhD (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); National Cancer Institute (NCI) (NIH); Sigma-Aldrich (Unknown)
Responsible Party: Sponsor-Investigator, Robert Bok, MD, PhD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22924; NCI-2022-09149 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); P41EB013598-11 (NIH); 5U01EB026412-04 (NIH); 5R01CA256740-02 (NIH)
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor
Keywords: Biomarker
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A / Phase 1: Feasibility Run-In (Experimental): Participants will undergo MR imaging at a single time point. Imaging will take one day and no follow up is planned.
  Interventions: Drug: Hyperpolarized 13C-Pyruvate; Procedure: Magnetic Resonance Imaging (MRI); Drug: 13C,15N-Urea
- Part B/ Phase II: Biomarker Cohort (Experimental): Participants will undergo paired 13C-pyruvate +/- 13C,15N-urea/metabolic MR imaging at baseline and again after approximately 21 days of therapy. Duration of the intervention period is approximately 21 days, and participants will be followed until discontinuation of their current SOC treatment regimen, about 6 months.
  Interventions: Drug: Hyperpolarized 13C-Pyruvate; Procedure: Magnetic Resonance Imaging (MRI); Drug: 13C,15N-Urea

INTERVENTIONS:
Drug: Hyperpolarized 13C-Pyruvate — Given IV
  Other Names: Hyperpolarized (HP) carbon^13 (13C)-pyruvate; HP-13C
Procedure: Magnetic Resonance Imaging (MRI) — Imaging procedure
  Other Names: MRI
Drug: 13C,15N-Urea — Given IV

SUMMARY:
This is a single center prospective imaging study investigating the utility of hyperpolarized 13C-pyruvate +/-13C,15N-Urea/ metabolic MR imaging. The current protocol will serve as a companion imaging biomarker study paired with standard of care (SOC) therapeutics, as well as investigational therapies that participants may be scheduled to receive outside of this protocol.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Phase I/Part A

1. To optimize the signal-to-noise ratio in detecting intra-tumoral hyperpolarized 13C pyruvate/lactate signal and hyperpolarized urea area under the curve (AUC) using metabolic magnetic resonance (MR) imaging in patients with advanced solid tumors.

Phase II/Part B

1. To determine the mean percent change from baseline in peak intra-tumoral hyperpolarized lactate-to-pyruvate ratio,pyruvate-to-lactate kinetic constant (kPL) and urea AUC after initiation of usual care/standard of care (SOC) treatment

SECONDARY OBJECTIVES:

Phase I/Part A

1. To further characterize the safety profile of hyperpolarized 13C-pyruvate +/- 13C,15N-urea.
2. To determine the reproducibility of intra-tumoral HP lac/pyr ratio with same-day repeated dose studies.

Phase II/Part B

1. To study the association between clinical outcomes and the percent change from baseline in peak intra-tumoral hyperpolarized lactate-to pyruvate ratio and kPL (+/-correction for HP urea AUC) after initiation of SOC treatment.
2. To further characterize the safety profile of hyperpolarized 13C pyruvate +/- 13C,15N-urea.
3. To determine the reproducibility of intra-tumoral HP lac/pyr ratio and/or HP urea AUC with same-day repeated dose studies.

OUTLINE:

Participants will be enrolled in Part A which is the feasibility, run-in study which includes the iterative adjustment of coil design to optimize imaging parameters within the target tumor lesion(s). If the data from Part A supports further investigation, additional participants will be enrolled in Part B which is a biomarker cohort which includes participants who are planning on being treated with either standard-of-care (SOC) or investigational therapies and will be followed until discontinuation of the treatment regimen outside of this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of at least one target pelvic, abdominal, thoracic, neck or extremity lesion detected by standard staging scans that, in the judgment of study investigator, would be amenable to hyperpolarized C-13 pyruvate/metabolic MR imaging:

   a. Target lesion must measure at least 1.0 cm in long axis diameter on Computerized tomography (CT) or magnetic resonance imaging (MRI).
2. The participant is able and willing to comply with study procedures and provide signed and dated informed consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
4. Adequate renal function defined as creatinine < 1.5 x upper limit of normal (ULN) or estimated creatinine clearance >50 mL/min (by the Cockcroft Gault equation).
5. Participants age 18 and older.

   Part B only:
6. Planned treatment for disease with either standard of care regimen or an investigational agent.

Exclusion Criteria:

1. Patients who because of age, general medical or psychiatric condition, or physiologic status cannot give valid informed consent.
2. Patients with contra- indications to MRI, such as cardiac pacemakers or non-compatible intracranial vascular clips.
3. Patients with a metallic implant or device that distorts local magnetic field and compromises the quality of MR imaging.
4. Patients with poorly controlled hypertension, defined as systolic blood pressure at study entry greater than 160mm Hg or diastolic blood pressure greater than 100mm Hg.

   Note: The addition of anti-hypertensives to control blood pressure is allowed.
5. Patients with congestive heart failure or New York Heart Association (NYHA) status >= 2.
6. Patients who are pregnant or lactating.
7. A history of clinically significant EKG abnormalities or myocardial infarction (MI) within 6 months of study entry.

   Note: Patients with rate-controlled atrial fibrillation/flutter will be allowed on study.
8. Any condition that, in the opinion of the Principal Investigator,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Signal-to-noise ratio (Part A) | Day of imaging (1 day)
  Signal-to-noise ratios is defined as a MR/spectroscopy parameter, consisting of the HP C13-Pyruvate or Lactate signal (peak) relative to background noise level (baseline) in MRI spectra of the tissue. For the analysis and interpretation of the HP 13C-pyruvate MR imaging data, DICOM software package (SIVIC) will be used to align, display and quantitatively interrogate serial multi-parametric imaging data.
Mean percent change from baseline in intratumoral HP pyruvate/lactate ratio | Up to 25 days
  Intra-tumoral region of interest (ROI) will be used to quantify peak HP lactate/pyruvate ratio values in the selected volumes of interest. Descriptive statistics will be used to characterize the mean change from baseline in intra-tumoral HP pyruvate/lactate ratio for the study cohort, along with a 95% confidence interval
Mean percent change from baseline in Urea Area Under Curve (AUC) | Up to 25 days
  Intra-tumoral region of interest (ROI) will be used to quantify urea AUC. Descriptive statistics will be used to characterize the mean change from baseline in Urea Area Under Curve (AUC)

SECONDARY OUTCOMES:
Number of participants reporting adverse events (Part A) | Day of imaging (1 day)
  Safety analyses will be performed for all patients having received a dose of HP 13C pyruvate HP 13C-pyruvate +/- 13C,15N-urea. Adverse events will be classified and graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE)
Number of participants reporting adverse events (Part B) | Up to 6 months
  Safety analyses will be performed for all patients having received a dose of HP 13C pyruvate HP 13C-pyruvate +/- 13C,15N-urea. Adverse events will be classified and graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE)
Median percent change from baseline in peak intratumoral hyperpolarized lactate-to-pyruvate ratio (Part B) | Up to 6 months
  Lactate/pyruvate ratio: hyperpolarized Lactate signal divided by the hyperpolarized pyruvate signal within the tumor region, for each injection/scan on the same day.
Median percent change from baseline in intra-tumoral HP Urea AUC (Part B) | Up to 6 months
  HP urea AUC within the tumor region, for each injection/scan on the same day
Objective response rate (ORR) (Part B) | Up to 6 months
  ORR is defined as the proportion of treated patients who experience an objective response (confirmed complete response (CR) or confirmed partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST)
Clinical benefit rate (CBR) (Part B) | Up to 6 months
  CBR is defined as the proportion of treated patients who experience clinical benefit (confirmed complete response (CR); confirmed partial response (PR); or stable disease (SD) for > 24 weeks per RECIST 1.1 criteria).
Radiographic progression-free survival (rPFS) (Part B) | Up to 6 months
  rPFS is defined as the amount of time that elapses between initiation of standard of care treatment and the day of first documented radiographic disease progression per RECIST v.1.1 or death from any cause.
Lactate/pyruvate ratio (Part B) | 1 day
  Intra-patient reproducibility of HP lac/pyr ratio and kPL for patients who undergo repeated dose imaging studies will be descriptively reported using summary statistics (mean difference, standard deviation, range).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bok, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No